CLINICAL TRIAL: NCT07260097
Title: Choroidal Venous Congestion Following Scleral Buckling - An Imaging Study
Acronym: SB
Status: Recruiting | Type: Observational
Sponsor: Singapore National Eye Centre (Other Government)
Responsible Party: Principal Investigator, Gemmy Cheung Chui Ming, Professor, Singapore National Eye Centre
Other Study IDs: 2025-0251
Record Dates: First submitted 2025-11-14; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Pachychoroid Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to understand how blood flow at the back of the eye changes over time after this surgery. By studying these changes, the investigators hope to gain insights that could help improve the understanding of other eye diseases, such as age-related macular degeneration (AMD) and polypoidal choroidal vasculopathy(PCV). This research may contribute to better treatments and outcomes for future patients.

DETAILED DESCRIPTION:
Scleral Buckling (SB) surgery emplaces a silicone band along the circumference of the eye to create an external support for retinal breaks, hence treating the retinal detachment. The investigators hypothesize that the presence of an external silicone band from the SB surgery would result in an increase in resistance across the choroidal venous outflow channels. This would in turn be manifested by quantitative and qualitative changes in choroidal vessel structure and architecture. These initial changes will eventually stabilise and revert to baseline after a period of long-term remodelling and adaptation.

Through this imaging study, the investigators aim to opportunistically study and validate these progressive choroidal vasculature changes in the choroidal outflow circulation following scleral buckle (SB) surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years and above
* Ability to provide informed consent
* First occurrence of a retinal detachment in one eye, deemed to require SB surgery with or without vitrectomy and/or cataract surgery.
* Clinically normal fellow eye (no previous intraocular surgery except for cataract extraction with lens implant, intraocular laser or injection procedures).

Exclusion Criteria:

* Affected eye undergoing vitreoretinal procedure other than an SB surgery with or without vitrectomy and/or cataract surgery.
* Pregnant or nursing women
* Persons who are unable to give informed consent

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 participants from the Singapore National Eye Centre.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-17 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Post operative choroidal venous congestion | 1 year
  Proportion of eyes demonstrating progression in choroidal venous congestion at 1 year, defined by increased choroidal thickness, increase in number of quadrants with pachyvessels, or new vortex vein anastomosis on multimodal imaging.

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore Eye Research Institute, Singapore, Singapore